CLINICAL TRIAL: NCT01558479
Title: The Parkinson's Genetic Research Study (PaGeR)
Brief Title: The Parkinson's Genetic Research Study
Acronym: PaGeR
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cyrus Zabetian, Professor of Neurology, University of Washington
Other Study IDs: 36777
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Genetics; Family Research; Hereditary Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Heredodegenerative Disorders, Nervous System

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood or saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Case: Has a diagnosis of Parkinson's disease
- Control: No diagnosis of Parkinson's disease
- Family Member: Has a family history of Parkinson's disease. Can be affected or unaffected with Parkinson's disease

SUMMARY:
The Parkinson's Genetic Research Study (PaGeR), headed by Dr. Cyrus Zabetian, is searching for genes that increase the risk of developing Parkinson's disease (PD) and related disorders. The study is a joint effort by neurologists and researchers across the United States and is sponsored by the National Institutes of Health. The coordinating center for PaGeR is located at the University of Washington and the VA Puget Sound Health Care System in Seattle.

DETAILED DESCRIPTION:
PaGeR is focusing on families in which two or more people have been diagnosed with PD. Past research suggests that such "multiplex" families might hold the key to the discovery of new PD genes.

To take part in PaGeR, participants will be asked to complete a questionnaire and to undergo an interview, a neurological exam, a short memory test, and a blood draw. Enrollment in the study usually takes between one and two hours. There is no cost to participate, and all study information is kept strictly confidential.

There are a number of designated sites across the country where families can enroll. However, for family members who are unable to travel to one of these sites, other arrangements can be made.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Member of a family in which there are two or more living individuals who have been diagnosed with Parkinson's disease

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families in which two or more people have been diagnosed with Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Zabetian, MD, MS, Principal Investigator — University of Washington, VA Puget Sound Health Care System
Locations (5):
- United States (5):
  - Emory University/ Wesley Woods Health Center, Atlanta, Georgia
  - University of Cincinnati, Cincinnati, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: Study Website — http://www.thepagerstudy.org